CLINICAL TRIAL: NCT06445465
Title: Phase 1 Study to Evaluate [18F]MNI-1216 ([18F]ACI-12589) as a Potential PET Radioligand for Imaging Alpha-synuclein Deposits in the Brain of Patients With Suspected Alpha-synuclein Pathology Compared With Healthy Volunteers
Brief Title: Study to Evaluate a Potential PET Radioligand for Imaging Alpha-synuclein Deposits in the Brain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Invicro (Other)
Collaborators: AC Immune SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9105
Record Dates: First submitted 2024-04-23; First posted 2024-06-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Alpha-Synucleinopathy; Parkinson's Disease; Dementia With Lewy Bodies; Multisystem Atrophy
MeSH Terms: conditions — Synucleinopathies; Parkinson Disease; Lewy Body Disease; Multiple System Atrophy

STUDY DESIGN:
Intervention Model Description: The study population will be composed of up to 30 subjects, including healthy volunteers and participants with α-synucleinopathies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with α-synucleinopathies. (Experimental): The study population will be composed of participants with α-synucleinopathies.
  Interventions: Drug: [18F]MNI-1216
- Healthy volunteers (Active Comparator): The study population will be composed of health volunteers.
  Interventions: Drug: [18F]MNI-1216

INTERVENTIONS:
Drug: [18F]MNI-1216 — [18F]MNI-1216 is an intravenously administered radioactive imaging agent being studied as a potential positron emitting radiopharmaceutical for in vivo imaging of α-synuclein deposits.
  Other Names: [18F]ACI-12589

SUMMARY:
The overall goal of this protocol is to evaluate [18F]MNI-1216 (also known as [18F]ACI-12589) as an α-synuclein targeted radiopharmaceutical in 3 parts as follows:

* Part 1: first in human (FiH) imaging
* Optional Part 2: expansion of FiH imaging
* Optional Part 3: retest imaging

A total of up to 30 participants may be enrolled and participate in the study. Part 1 of the study will include up to 10 participants (target of up to 5 healthy volunteers and up to 5 participants with idiopathic Parkinson's Disease). There will be an ongoing review of study data in Part 1 to evaluate the characteristics of tracer binding and safety. If the study results are deemed adequate in Part 1, Part 2 and/or Part 3 may be initiated. The decision to initiate Part 3 may also include a review of data from Part 2, if Part 2 is performed and the data are available. If performed, Part 2 will include up to 20 participants, including health volunteers and participants with α-synucleinopathies to acquire additional tracer-related data. If performed, Part 3 will include up to 10 participants from in Part 1 and/or Part 2 (including health volunteers and participants with α-synucleinopathies) to evaluate the reliability of [18F]MNI-1216 ([18F]ACI-12589) Positron Emission Tomography (PET) imaging.

DETAILED DESCRIPTION:
The overall goal of this protocol is to evaluate [18F]MNI-1216 (also known as [18F]ACI-12589) as an α-synuclein targeted radiopharmaceutical in 3 parts.

The specific objective for Parts 1, 2, and 3 is:

• To characterize [18F]MNI-1216 ([18F]ACI-12589) as a PET radioligand for imaging α-synuclein pathology.

The additional specific objectives for Part 1 and Part 2 are:

* To visually and quantitatively assess brain uptake and pharmacokinetics of [18F]MNI-1216 ([18F]ACI-12589) as a PET imaging marker for α-synuclein pathology in individuals with α-synucleinopathies (including idiopathic PD) compared with corresponding data from healthy volunteer participants.
* To evaluate the safety of a single injection of [18F]MNI-1216 ([18F]ACI-12589).

The additional specific objectives for Part 3 are:

* To evaluate the reliability (test/retest) of [18F]MNI-1216 ([18F]ACI-12589) parameters in individuals with α-synucleinopathies and healthy volunteers.
* To evaluate the safety of up to 2 injections of [18F]MNI-1216 ([18F]ACI-12589).

For each subject participating in the study, the duration of study participation will be up to 78 days.

In Part 1 and Part 2 (if Part 2 is performed), screening assessments will occur within 30 days prior to the Baseline [18F]MNI-1216 ([18F]ACI-12589) Imaging Visit (Day 1). If determined to be necessary by the study team, subjects may participate in an [18F]Florbetapir Imaging Visit up to 6 weeks following Day 1 (will be completed between Day 2 and Day 42). A Safety Phone Call for adverse event assessment will occur 4 days (±2 days) following each imaging visit performed. In Part 3 (if performed), subjects will participate in a Retest [18F]MNI-1216 ([18F]ACI-12589) Imaging Visit between Day 4 and Day 29 (within 3 days to 4 weeks) following the Baseline [18F]MNI-1216 ([18F]ACI-12589) Imaging Visit (Day 1). A Safety Phone Call for adverse event assessment will occur 4 days (±2 days) following the retest imaging visit, if performed.

ELIGIBILITY:
Inclusion Criteria:

* Participants is able to provide written informed consent, which must be obtained before any assessment is performed.
* Female participants must not be of childbearing potential, or agree to use contraception and not donate eggs if of childbearing potential. At the discretion of the Investigator, participants without documentation of non-childbearing potential may receive pregnancy testing.

  * A woman is considered to be of childbearing potential if postmenarchal, has not reached a postmenopausal state (12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (ie, removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the PI (eg, Müllerian agenesis).
  * Women of childbearing potential must commit to remain abstinent (refrain from heterosexual intercourse) or use 2 forms of birth control, 1 of which is a barrier contraception method, for the duration of the study and 30 days after study completion. Periodic abstinence (eg, calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
  * Women of childbearing potential must commit to not donate ovum for the duration of the study and 30 days after study completion.
* Male participants and their partners of childbearing potential must commit to the use of 2 methods of contraception, 1 of which is a barrier method for male participants for the study duration and 90 days after study completion.
* Male participants must not donate sperm for the study duration and for 90 days after study completion.
* Willing and able to cooperate with study procedures.
* For participants receiving arterial cannulation, adequate circulation to the hand for safe placement of arterial line (as determined by Allen's test) and blood clotting (PT and PTT).
* If participant takes bupropion, participant must agree to hold this medication for at least 12 hours prior to DaTscan imaging (if performed).

Additional Inclusion Criteria for healthy volunteers:

* Males and females aged ≥ 21 years.
* Healthy with no clinically relevant finding on physical examination at Screening and upon reporting to the clinic for the [18F]MNI-1216 ([18F]ACI-12589) Imaging Visit.
* No family history of α-synucleinopathy, including PD, or other early-onset neurological disease associated with dementia.
* No personal history of clinically significant neurologic and/or psychiatric disorders.
* No evidence of dopamine transporter deficit on DaTscan performed either as part of Screening or on previously acquired DaTscan (within 6 months prior to signing consent).
* Have a Montreal Cognitive Assessment (MoCA) score ≥ 26.
* No cognitive impairment as judged by the PI.

Additional Inclusion Criteria for Participants with α-synucleinopathy:

* Males and females aged ≥ 40 years.
* Participants diagnosed with any of the following:

  * Idiopathic Parkinson's Disease
  * Parkinson's Disease with genetic risk factor (except leucine-rich repeat kinase 2 [LRRK2] mutation)
  * Dementia with Lewy Bodies
  * Multisystem Atrophy
* A brain MRI consistent with a diagnosis of α-synucleinopathy, with no evidence of focal disease to account for the participant's neurological symptoms or MRI exclusion criteria listed below under "Exclusion Criteria".
* Evidence of dopamine transporter deficit on DaTscan performed either as part of Screening or on previously acquired DaTscan.
* Medications taken for symptomatic treatment of α-synucleinopathy must be maintained on a stable dosage regimen for at least 30 days before Screening Visit.
* Ability to tolerate lying in the scanner for up to ~180 minutes without excessive head or jaw tremor or dyskinesia sufficient to cause significant motion artifact on the PET scans.

Exclusion Criteria:

* Current or prior history of any alcohol or drug abuse in the past 2 years.
* Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness.
* Known history of hypersensitivity, including hypersensitivity to the active substances used for DaTscan, [18F]MNI-1216 ([18F]ACI-12589) and [18F]florbetapir or derivatives, or to any of the associated excipients.
* Participant has received an investigational drug within 30 days or five half-lives prior to the baseline assessments, whichever is longer.
* Prior participation in other research protocols or clinical care during the past year that would result in radiation exposure to an effective radiation dose exceeding the acceptable annual limit established by the US Federal Guidelines (effective dose of 50 mSv, including the procedures in this clinical protocol).
* Pregnant, lactating or breastfeeding.
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Unsuitable veins for repeated venipuncture.
* MRI with clinically significant structural abnormalities.
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, central nervous system (CNS) aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.
* Participant has received treatment with a drug, antibody or vaccine targeting α-synuclein.
* Ongoing treatment with methylphenidate, modafinil, metoclopramide, alpha methyldopa, reserpine, or amphetamine derivative is prohibited 24 hours or during a period corresponding to 5 half-lives of the compound, whichever longer, prior to DaTscan imaging.
* Treatment with any antihemostasis medication (eg, warfarin, heparin, thrombin inhibitors, Factor Xa inhibitors, streptokinase, urokinase, tissue plasminogen activators) within 2 weeks of the planned arterial cannula placement (if performed) for either the baseline or retest imaging.

Additional Exclusion Criteria for Participants with α-synucleinopathy:

* Evidence of early frequent falls or eye movement abnormalities consistent with PSP.
* Individuals with known LRRK2 mutation (based on previous source documentation).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Volume of distribution (VT) of [18F]MNI-1216 across multiple brain regions | up to 78 days
  Volume of distribution (VT) across multiple brain regions will be measured and comparison between participants with α-synucleinopathies and healthy volunteers will be performed to visually and quantitatively assess brain uptake and pharmacokinetics of [18F]MNI-1216 ([18F]ACI-12589) as a PET imaging marker for α-synuclein pathology in individuals with α-synucleinopathies.
Number of participants with [18F]MNI-1216-related adverse events as assessed by CTCAE | up to 78 days
  Participants will be monitored to evaluate the safety of a single injection of [18F]MNI-1216 ([18F]ACI-12589). The following assessments will be performed to monitor participants for adverse reactions:
  * Clinical laboratory tests.
  * Vital signs.
  * Physical findings.
  * Electrocardiograms

OTHER OUTCOMES:
Average variability across subjects | up to 78 days
  To evaluate the reliability (test/retest) of parameters in individuals with α-synucleinopathies and healthy volunteers, Investigators will calculate the average and standard deviation of variability across subjects based on imaging data ((test - retest) / average (test, retest)).
Intraclass correlation (ICC) of test and retest scans | up to 78 days
  To evaluate the reliability (test/retest) of parameters in individuals with α-synucleinopathies and healthy volunteers, Investigators will calculate the intraclass correlation of test and retest scans from imaging data. Intraclass correlation is a reliability index in test/retest analyses.

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, MD, Principal Investigator — Invicro
Locations (1):
- Invicro, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No